CLINICAL TRIAL: NCT02786485
Title: A Phase I Study of Matched Unrelated Donor BPX-501 T Cell Infusion for Adults With Recurrent or Minimal Residual Disease Hematologic Malignancies Post-Allogeneic Transplant
Brief Title: Study of Matched Unrelated Donor T Cell Infusion for Hematologic Malignancies After Allo-HSCT
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Bellicum Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP-008-MUD
Expanded Access: NCT03639844 (No longer available)
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Lymphomas; Multiple Myeloma; Other High-risk Hematological Malignancies
Keywords: BPX-501; Rimiducid; AP1903; Hematological malignancies; Hematologic diseases; Leukemias and Myelodysplastic Syndromes; Lymphomas; Multiple myeloma
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Lymphoma; Multiple Myeloma; Hematologic Neoplasms; Hematologic Diseases | interventions — AP 1903 reagent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rivogenlecleucel & Rimiducid (Experimental): All subjects will receive 3 courses of rivogenlecleucel (BPX-501 T cells) infusions at 30 day intervals with 2 escalating dose levels (DL). DL1 on Day 0 and DL2 on Days 30 and 60.
  Escalating doses of rimiducid (AP1903) (0.1 mg/kg and 0.4 mg/kg) will be investigated for the treatment of aGvHD after rivogenlecleucel infusion.
  Interventions: Biological: rivogenlecleucel; Drug: Rimiducid

INTERVENTIONS:
Biological: rivogenlecleucel — T cells transduced with iCasp safety switch
  Other Names: BPX-501
Drug: Rimiducid — administered to treat GVHD
  Other Names: AP1903

SUMMARY:
This is a Phase I, multicenter, open-label, non-randomized study of matched unrelated donor BPX-501 T cell infusion in adult subjects with hematological malignancies presenting with recurrent disease minimal residual disease (MRD) post-allogeneic transplant.

DETAILED DESCRIPTION:
Un-manipulated donor lymphocyte infusion (DLI) is used after stem cell transplantation to treat and prevent relapse, to prevent infections and to establish full donor chimerism. The addition of mature T cells which exhibit a broad repertoire of T cell immunity against viral antigens, as well as against cancer antigens, might provide a clinical benefit. However, an expected side effect of the presence of mature T cells is the potential occurrence of acute graft-versus-host disease (aGvHD). The use of a suicide gene switch which would trigger the initiation of the apoptosis of the alloreactive T cells by the infusion of a drug would represent the potential optimal strategy for restoring early immunity with a built in "safety switch" against GvHD side effects. Evidence has emerged that low-dose DLI followed by dose escalation can achieve higher clinical response rate with lower GvHD occurrence. Optimization of DLI dose and schedule as well as strategies of donor T-cell manipulation may lead to the consistent ability to separate GvHD from graft-versus-tumor (GvT) activity and improve the safety of DLI treatment. Our strategy is to infuse escalating doses of manipulated T cells (from the same donor who provided the original hematopoietic stem cell graft) in adults and children with recurrent or minimal residual disease (MRD) hematologic malignancies post-allogeneic transplant to accelerate immune reconstitution thus improving graft versus leukemic effect while reducing the severity of GvHD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥ 18 yrs and ≤ 65 yrs;
* Clinical diagnosis of one of the following hematological malignancies:

  * Leukemia
  * Myelodysplastic Syndromes
  * Lymphomas
  * Multiple Myeloma
  * Other high-risk hematological malignancy eligible for stem cell transplantation per institutional standard;
* Recurrent disease that presents ≥100 days after, or minimal residual disease (MRD) that presents ≥ 30 days following a hematopoietic stem cell transplant (HSCT) using a matched unrelated donor located through the National Marrow Donor Program (NMDP);
* Life expectancy >10 weeks;
* Signed donor and patient/guardian informed consent;
* A 8/8 genotypic identical match as determined by high resolution typing for the following genetic loci: human leukocyte antigen (HLA)-A, HLA-B, HLA-C and HLA-DRB1;
* Performance status: Karnofsky score > 50%;
* Subjects with adequate organ function as measured by:

  * Bone marrow:

    * > 25% donor T-cell chimerism post-transplant
    * Absolute neutrophil count (ANC) >1 x 109/L
  * Cardiac: left ventricular ejection fraction (LVEF) at rest ≥ 45%
  * Pulmonary: forced expiratory volume (FEV) 1, forced vital capacity (FVC), diffusion capacity of lunch for carbon monoxide (DLCO) ≥ 50% predicted (corrected for hemoglobin)
  * Hepatic: direct bilirubin ≤ 3x upper limit of normal (ULN), or aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 5x ULN
  * Renal: creatinine ≤ 2x of ULN for age.

Exclusion Criteria:

* ≥ Grade II acute GVHD or chronic extensive GVHD due to a previous allograft at the time of screening;
* Active central nervous system (CNS) involvement with malignant cells (≤ 2 months prior to consenting);
* Current uncontrolled bacterial, viral or fungal infection (currently taking medication with evidence of progression of clinical symptoms or radiologic findings); the principal investigator is the final arbiter of this criterion;
* Positive HIV serology or viral RNA;
* Pregnancy (positive serum β human chorionic gonadotropin [HCG] test) or breast-feeding;
* Fertile men or women unwilling to use effective forms of birth control or abstinence for one year after transplantation;
* Bovine product allergy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Adverse events | 30 days after last dose of study drug (BPX-501 and/or rimiducid)
  Number of adverse events after study drug (BPX-501 and/or rimiducid) administration as a measure of safety

CONTACTS AND LOCATIONS:
Overall Officials: Bellicum Pharmaceuticals, Study Director — Bellicum Pharmaceuticals, Inc.

IPD SHARING:
Plan to Share IPD: No